CLINICAL TRIAL: NCT03191604
Title: A Multicenter Study Evaluating the Impact of NBI on Patients With Barrett's Esophagus Associated Neoplasia Undergoing Endoscopic Eradication Therapy (EET)
Brief Title: Impact of NBI on Patients Undergoing Endoscopic Eradication Therapy
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sri Komanduri, Director of Endoscopy, Northwestern University
Other Study IDs: STU00205021
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Barrett Esophagus
Keywords: Endoscopy; Narrow band imaging; Dysplasia
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopists familiar with EET: Physicians familiar with conducting endoscopic eradication therapy.
  Interventions: Other: Video intervention

INTERVENTIONS:
Other: Video intervention — Video clips of endoscopy footage with just HD-WLE and clips with NBI will be shown to endoscopists.

SUMMARY:
This study tests the impact of narrow band imaging (NBI) on endoscopists' accurate detection of visible lesions and dysplasia in patients with Barrett's esophagus, as well as the effect of NBI on the choice of primary treatment modality among endoscopists performing endoscopic eradication therapy (EET).

DETAILED DESCRIPTION:
Barrett's esophagus (BE), is a condition whereby normal esophageal squamous epithelium is replaced by metaplastic columnar epithelium, predisposing patients to esophageal adenocarcinoma (EAC). It is estimated that about 5.6% of adults in the United States have BE with risk factors including: long standing gastroesophageal reflux disease, tobacco use, male gender, central obesity, and age over 50 years. EAC is believed to progress in a step-wise pattern with the following order of non-dysplastic BE, low-grade dysplasia (LGD), and high-grade dysplasia (HGD). Each carries a risk of progression to EAC, differing by degree of dysplasia: 0.2-0.5%, 0.7%, and 7% per year, respectively. Given this association, it is common practice to perform endoscopic surveillance with biopsies in patients with BE. Endoscopic surveillance has been shown to detect EAC at earlier stages and improve survival in asymptomatic presentations. As dysplasia in BE may not always be seen as a distinct lesion, surveillance programs entail use of the Seattle Protocol, a systematic four-quadrant biopsy technique obtained at 1 to 2 cm increments. Current guidelines recommend the use of high-definition white light endoscopy (HD-WLE) as it is superior over standard-definition in regards to improved targeted detection of dysplasia.

Advanced endoscopic imaging techniques have been proposed to improve dysplasia detection with preference for electronic chromoendoscopy, specifically narrow band imaging (NBI), as it does not require dye sprays. NBI has been shown to be more accurate in detecting intestinal metaplasia and HGD. HGD is more often detected in areas with subtle mucosal and vascular abnormalities, which may be more difficult to see on HD-WLE alone. However, subtle lesions may go undetected, as NBI is not routinely used in the community with a recent survey showing only about a third of practicing gastroenterologists use advanced endoscopic imaging. The widespread use of NBI has been potentially limited by a perceived complexity of interpretation and lack of standardization. Recently, Sharma et al introduced the BING criteria - a standardized classification system to detect dysplasia and EAC with NBI. While a few studies have demonstrated no significant difference in detection of dysplasia or neoplasia between HD-WLE and NBI, they have had some limitations. The studies occurred prior to the BING classification system, and participants were limited to a few expert tertiary medical centers.

The current standard of care for visible lesions identified by HD-WLE (nodules, ulcers, erosions, or plaques) is endoscopic mucosal resection (EMR). Endoscopic recognition and appropriate resection of visible lesions is essential for optimal patient outcomes. Staging EMR is critical as it allows for histopathological "upgrading" or "downgrading" of dysplasia and ultimately is the best tool for identifying and treating early EAC. Despite the importance of EMR for BE-AN, survey data suggests it is underutilized in practice with 39% of academic endoscopists and 13% of community-based endoscopists performing EMR. While many endoscopists utilize NBI to assist in identification of visible lesions, the resection of areas deemed "abnormal" by NBI alone is not widely accepted. Moreover, endoscopists at community hospitals detect neoplastic lesions at significantly lower rates than at BE expert centers.

Given these data, routine use of NBI prior to EET could significantly impact treatment decisions among all endoscopists with highly accurate rates of dysplasia detection. It's been shown that NBI increases the accuracy and positive predictive value of predicting histology than if HD-WLE is used alone. This study is limited by the use of still-images, which does not accurately reproduce live images seen during endoscopy. Nevertheless, the current standard of using HD-WLE for identification of visible lesions likely underestimates the presence of dysplastic areas in patients undergoing Endoscopic Eradication Therapy (EET) for BE-AN. We hypothesize that the routine use of narrow band imaging (NBI) for identification of visible lesions will improve dysplasia detection and have a significant effect on the choice of primary treatment modality among endoscopists performing EET. To this end, we propose a video-based study to evaluate the impact of NBI on choice of treatment modality during EET.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists familiar with EET.

Exclusion Criteria:

* Endoscopists not familiar with EET or non-endoscopists.
* Special populations will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endoscopist sub-groups include academic endoscopists performing greater than 50 EET procedures per year, community endoscopists performing greater than 50 EET procedures per year, 25 academic gastroenterologists performing greater than 500 upper endoscopies per year not including EET, and 25 community gastroenterologists performing greater than 500 upper endoscopies per year not including EET.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Altered chosen treatment modality due to NBI | 1 year
  Percentage of cases in which use of NBI altered decision-making in regards to initial treatment modality for patients undergoing EET.

SECONDARY OUTCOMES:
% visable dysplastic lesions detected | 1 year
  Percentage of visible dysplastic lesions detected by HD-WLE and NBI across all participants stratified by subgroup of experience
Accurate pathology assessment | 1 year
  Accuracy of pathology assessment by endoscopists using HD-WLE and NBI in patients undergoing EMR
Differences in pathology identification between subgroups | 1 year
  Differences in identification of pathology based on subgroup of experience, volume of EET, and type of practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spechler SJ, Souza RF. Barrett's esophagus. N Engl J Med. 2014 Aug 28;371(9):836-45. doi: 10.1056/NEJMra1314704. No abstract available. PMID 25162890
- [Background] Hayeck TJ, Kong CY, Spechler SJ, Gazelle GS, Hur C. The prevalence of Barrett's esophagus in the US: estimates from a simulation model confirmed by SEER data. Dis Esophagus. 2010 Aug;23(6):451-7. doi: 10.1111/j.1442-2050.2010.01054.x. Epub 2010 Mar 26. PMID 20353441
- [Background] Ireland CJ, Thompson SK, Laws TA, Esterman A. Risk factors for Barrett's esophagus: a scoping review. Cancer Causes Control. 2016 Mar;27(3):301-23. doi: 10.1007/s10552-015-0710-5. Epub 2016 Feb 5. PMID 26847374
- [Background] Shaheen NJ, Falk GW, Iyer PG, Gerson LB; American College of Gastroenterology. ACG Clinical Guideline: Diagnosis and Management of Barrett's Esophagus. Am J Gastroenterol. 2016 Jan;111(1):30-50; quiz 51. doi: 10.1038/ajg.2015.322. Epub 2015 Nov 3. PMID 26526079
- [Background] Incarbone R, Bonavina L, Saino G, Bona D, Peracchia A. Outcome of esophageal adenocarcinoma detected during endoscopic biopsy surveillance for Barrett's esophagus. Surg Endosc. 2002 Feb;16(2):263-6. doi: 10.1007/s00464-001-8161-3. Epub 2001 Nov 16. PMID 11967675
- [Background] Ferguson MK, Durkin A. Long-term survival after esophagectomy for Barrett's adenocarcinoma in endoscopically surveyed and nonsurveyed patients. J Gastrointest Surg. 2002 Jan-Feb;6(1):29-35; discussion 36. doi: 10.1016/s1091-255x(01)00052-x. PMID 11986015
- [Background] Fountoulakis A, Zafirellis KD, Dolan K, Dexter SP, Martin IG, Sue-Ling HM. Effect of surveillance of Barrett's oesophagus on the clinical outcome of oesophageal cancer. Br J Surg. 2004 Aug;91(8):997-1003. doi: 10.1002/bjs.4591. PMID 15286961
- [Background] van Sandick JW, van Lanschot JJ, Kuiken BW, Tytgat GN, Offerhaus GJ, Obertop H. Impact of endoscopic biopsy surveillance of Barrett's oesophagus on pathological stage and clinical outcome of Barrett's carcinoma. Gut. 1998 Aug;43(2):216-22. doi: 10.1136/gut.43.2.216. PMID 10189847
- [Background] Fitzgerald RC, Saeed IT, Khoo D, Farthing MJ, Burnham WR. Rigorous surveillance protocol increases detection of curable cancers associated with Barrett's esophagus. Dig Dis Sci. 2001 Sep;46(9):1892-8. doi: 10.1023/a:1010678913481. PMID 11575441
- [Background] Abela JE, Going JJ, Mackenzie JF, McKernan M, O'Mahoney S, Stuart RC. Systematic four-quadrant biopsy detects Barrett's dysplasia in more patients than nonsystematic biopsy. Am J Gastroenterol. 2008 Apr;103(4):850-5. doi: 10.1111/j.1572-0241.2007.01746.x. Epub 2008 Mar 26. PMID 18371135
- [Background] Sami SS, Subramanian V, Butt WM, Bejkar G, Coleman J, Mannath J, Ragunath K. High definition versus standard definition white light endoscopy for detecting dysplasia in patients with Barrett's esophagus. Dis Esophagus. 2015 Nov-Dec;28(8):742-9. doi: 10.1111/dote.12283. Epub 2014 Sep 10. PMID 25209721
- [Background] Song J, Zhang J, Wang J, Guo X, Yu S, Wang J, Liu Y, Dong W. Meta-analysis of the effects of endoscopy with narrow band imaging in detecting dysplasia in Barrett's esophagus. Dis Esophagus. 2015 Aug-Sep;28(6):560-6. doi: 10.1111/dote.12222. Epub 2014 Apr 24. PMID 24758693
- [Background] Jayasekera C, Taylor AC, Desmond PV, Macrae F, Williams R. Added value of narrow band imaging and confocal laser endomicroscopy in detecting Barrett's esophagus neoplasia. Endoscopy. 2012 Dec;44(12):1089-95. doi: 10.1055/s-0032-1325734. Epub 2012 Nov 27. PMID 23188660
- [Background] Singh M, Gupta N, Gaddam S, Balasubramanian G, Wani S, Sinh P, Aghaie K, Higbee AD, Rastogi A, Kanakadandi V, Bansal A, Sharma P. Practice patterns among U.S. gastroenterologists regarding endoscopic management of Barrett's esophagus. Gastrointest Endosc. 2013 Nov;78(5):689-95. doi: 10.1016/j.gie.2013.05.002. Epub 2013 Jun 14. PMID 23769458
- [Background] Sharma P, Bergman JJ, Goda K, Kato M, Messmann H, Alsop BR, Gupta N, Vennalaganti P, Hall M, Konda V, Koons A, Penner O, Goldblum JR, Waxman I. Development and Validation of a Classification System to Identify High-Grade Dysplasia and Esophageal Adenocarcinoma in Barrett's Esophagus Using Narrow-Band Imaging. Gastroenterology. 2016 Mar;150(3):591-8. doi: 10.1053/j.gastro.2015.11.037. Epub 2015 Nov 25. PMID 26627609
- [Background] Sharma P, Hawes RH, Bansal A, Gupta N, Curvers W, Rastogi A, Singh M, Hall M, Mathur SC, Wani SB, Hoffman B, Gaddam S, Fockens P, Bergman JJ. Standard endoscopy with random biopsies versus narrow band imaging targeted biopsies in Barrett's oesophagus: a prospective, international, randomised controlled trial. Gut. 2013 Jan;62(1):15-21. doi: 10.1136/gutjnl-2011-300962. Epub 2012 Feb 7. PMID 22315471
- [Background] Scholvinck DW, van der Meulen K, Bergman JJGHM, Weusten BLAM. Detection of lesions in dysplastic Barrett's esophagus by community and expert endoscopists. Endoscopy. 2017 Feb;49(2):113-120. doi: 10.1055/s-0042-118312. Epub 2016 Nov 17. PMID 27855466
- [Background] Singh R, Jayanna M, Wong J, Lim LG, Zhang J, Lv J, Liu D, Lee YC, Han ML, Tseng PH, Namasivayam V, Banerjee R, Uedo N, Chan WK, Ho SH, Chen SY, Bhatia S, Funasaka K, Ando T, Wu J, Lesmana C, Tam W, Wang WL, Chang CY, Jung HY, Jung KW, Bestari MB, Yao K, Chong VH, Sharma P, Ho KY. Narrow-band imaging and white-light endoscopy with optical magnification in the diagnosis of dysplasia in Barrett's esophagus: results of the Asia-Pacific Barrett's Consortium. Endosc Int Open. 2015 Feb;3(1):E14-8. doi: 10.1055/s-0034-1377610. Epub 2014 Sep 26. PMID 26134765